CLINICAL TRIAL: NCT04109599
Title: A Digital Intervention to Prevent the Initiation of Opioid Misuse in Adolescents in School-based Health Centers
Brief Title: A Digital Intervention to Prevent Initiation of Opioid Misuse in Adolescents in School-based Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000026247; 1UG3DA050251-01 (NIH)
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Opioid Misuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- PlaySmart Full Game (Experimental): Adolescents, boys and girls, aged 16-19 participated in the pilot testing of the adapted game. PlaySmart is a digital intervention targeted towards preventing opioid misuse in older adolescents.
  Interventions: Behavioral: PlaySmart
- Trading Wisdom Storyline (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player receives an opioid prescription from their dentist. This storyline includes information about safe use of opioids and the difference between use and misuse.
  Interventions: Behavioral: PlaySmart Storyline
- Lean on Me Storyline (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player is offered opioids at a party. This storyline includes information about different forms of opioids and their effects.
  Interventions: Behavioral: PlaySmart Storyline
- Tough Love Storyline (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player navigates supporting their partner struggling with opioid misuse. This storyline includes information about treatment and recovery resources for opioid misuse & Opioid Use Disorder.
  Interventions: Behavioral: PlaySmart Storyline
- Grandma's Pills Storyline (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player witnesses the sharing of an opioid prescription within their family. This storyline includes information about medication safety and opioid overdose identification and response.
  Interventions: Behavioral: PlaySmart Storyline
- A Friend in Need Storyline (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player interacts with a friend that is in distress. This storyline includes information about how to navigate peer-to-peer support.
  Interventions: Behavioral: PlaySmart Storyline
- A New Direction Storyline (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player seeks out therapy as an option to manage stress. This storyline includes information about how to seek professional help for mental health.
  Interventions: Behavioral: PlaySmart Storyline
- Risk Sense All Levels (Experimental): Adolescents, boys and girls, aged 16-19 participated in beta testing all levels of this PlaySmart mini game intended to increase perceived risk of harm of opioid misuse.
  Interventions: Behavioral: Play Smart Mini-Game
- PlaySmart Full Game: Focus on Character Development (Experimental): Adolescents, boys and girls, aged 16-19 participated in the pilot testing of the adapted game. PlaySmart is a digital intervention targeted towards preventing opioid misuse in older adolescents. Participants in this arm focused on beta testing character development aspects throughout the game.
  Interventions: Behavioral: PlaySmart

INTERVENTIONS:
Behavioral: PlaySmart — Participants played the developed PlaySmart game over the course of a week.
  Arms: PlaySmart Full Game; PlaySmart Full Game: Focus on Character Development
Behavioral: PlaySmart Storyline — Participants played through one PlaySmart Storyline during one 1-1.5 hour session.
  Arms: A Friend in Need Storyline; A New Direction Storyline; Grandma's Pills Storyline; Lean on Me Storyline; Tough Love Storyline; Trading Wisdom Storyline
Behavioral: Play Smart Mini-Game — Participants played through all levels of the PlaySmart Risk Sense mini-game during one 1-1.5 hour session.
  Arms: Risk Sense All Levels

SUMMARY:
This study's specific aims were to: develop a digital intervention as a prevention intervention through focus groups with 40 youth; pilot-test the developed digital intervention with 30 adolescents, using methods from the investigator's prior research; develop implementation strategies and partners through focus groups with 50 School Based Health Alliance affiliates and 30 adolescents from an Advisory Council.

DETAILED DESCRIPTION:
Most opioid misuse begins during adolescence and young adulthood. Adolescence is the time to intervene with prevention interventions (i.e., interventions focused on adolescents who have not yet misused opioids) in settings like school-based health centers (HCs), yet few interventions exist that prevent initiation of opioid misuse. "Serious videogame" interventions can improve health behaviors. They meet adolescents "where they are," and compared to standard interventions, they can reach large populations, with consistent fidelity, place limited demands on personnel/resources, and facilitate rapid sustainable distribution, all at a potentially lower cost.

This study harnessed the power of videogame interventions and incorporated components of effective substance use prevention programs to develop an evidence-informed intervention to prevent the initiation of opioid misuse in adolescents. Building on our experience developing videogame interventions and in partnership with the national School-Based Health Alliance (SBHA), we developed and tested a new videogame intervention, PlaySmart.

PlaySmart was built upon our PlayForward videogame intervention platform that has demonstrated efficacy in improving attitudes and knowledge related to risk behaviors. Through rigorous formative work and with input from adolescents, and our SBHA and game development partners, we created the PlaySmart videogame intervention.

PlaySmart is designed to provide players with behavioral skills and knowledge through repetitive and engaging videogame play to target adolescent perception of risk of harm from initiating opioid misuse.

The gap in the research on preventing initiation of opioid misuse in youth and in implementing prevention programs with good fidelity needs to be urgently addressed given the high prevalence of adolescent opioid misuse and overdose. This research has the potential to create a videogame intervention to prevent initiation of opioid misuse with far-reaching and sustained impact on adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent participants must attend high school that has a school-based health center, to participate in pilot testing

Exclusion Criteria:

* Failure to meet Inclusion Criteria

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Fiellin, MD, Principal Investigator — Director, play2PREVENT Lab at Yale, Internal Medicine
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: PlaySmart Full Game: Adolescents, boys and girls, aged 16-19 participated in the pilot testing of the adapted game. PlaySmart is a digital intervention targeted towards preventing opioid misuse in older adolescents.
- Experimental: Trading Wisdom Storyline: Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player receives an opioid prescription from their dentist. This storyline includes information about safe use of opioids and the difference between use and misuse.
- Experimental: Lean on Me Storyline: Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player is offered opioids at a party. This storyline includes information about different forms of opioids and their effects.
- Experimental: Tough Love Storyline: Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player navigates supporting their partner struggling with opioid misuse. This storyline includes information about treatment and recovery resources for opioid misuse & Opioid Use Disorder
- Experimental: Grandma's Pills Storyline: Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player witnesses the sharing of an opioid prescription within their family. This storyline includes information about medication safety and opioid overdose identification and response.
- Experimental: A Friend in Need Storyline: Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player interacts with a friend that is in distress. This storyline includes information about how to navigate peer-to-peer support.
- Experimental: A New Direction Storyline: Adolescents, boys and girls, aged 16-19 participated in beta testing this PlaySmart storyline where the player seeks out therapy as an option to manage stress. This storyline includes information about how to seek professional help for mental health.
- Experimental: Risk Sense All Levels: Adolescents, boys and girls, aged 16-19 participated in beta testing all levels of this PlaySmart mini game intended to increase perceived risk of harm of opioid misuse.
- Experimental: PlaySmart Full Game: Focus on Character Development: Adolescents, boys and girls, aged 16-19 participated in the pilot testing of the adapted game. PlaySmart is a digital intervention targeted towards preventing opioid misuse in older adolescents. Participants in this arm focused on beta testing character development aspects throughout the game.
Period: Overall Study
Arm/Group | Experimental: PlaySmart Full Game | Experimental: Trading Wisdom Storyline | Experimental: Lean on Me Storyline | Experimental: Tough Love Storyline | Experimental: Grandma's Pills Storyline | Experimental: A Friend in Need Storyline | Experimental: A New Direction Storyline | Experimental: Risk Sense All Levels | Experimental: PlaySmart Full Game: Focus on Character Development
Started | 3 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3
Completed | 3 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were collected prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: PlaySmart Full Game | Experimental: Trading Wisdom Storyline | Experimental: Lean on Me Storyline | Experimental: Tough Love Storyline | Experimental: Grandma's Pills Storyline | Experimental: A Friend in Need Storyline | Experimental: A New Direction Storyline | Experimental: Risk Sense All Levels | Experimental: PlaySmart Full Game: Focus on Character Development | Total
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 33
Age, Customized [Mean (Full Range); unit: years] | 17 [17 to 17] | 17 [16 to 18] | 16.5 [16 to 18] | 16.5 [16 to 17] | 16.5 [16 to 17] | 17.25 [17 to 18] | 17 [16 to 19] | 16.6 [16 to 18] | 17 [17 to 17] | 16.8 [16 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 3 | 3 | 3 | 4 | 1 | 1 | 21
  Male | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 6
  Not Hispanic or Latino | 3 | 2 | 4 | 4 | 4 | 2 | 4 | 1 | 2 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 1 | 4 | 2 | 1 | 1 | 0 | 14
  White | 0 | 4 | 2 | 2 | 0 | 0 | 2 | 0 | 1 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 33
Knowledge Questions [Mean (Standard Deviation); unit: Percentage of Questions Correct] — Population: Knowledge questions included 5 true/false questions about opioid misuse. Only the "PlaySmart Full Game" arm (n=3) was asked knowledge questions at baseline and post gameplay. Qualitative focus group feedback was collected from all other arms.
  Percentage of Questions Correct
    number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    (all) | 80 (0) |  |  |  |  |  |  |  |  | 80 (0)
Perception of Risk of Harm Questions [Mean (Full Range); unit: units on a scale] — Population: Participants were asked 5 perception of harm questions and then asked to rate the questions on a 4-point scale (no risk to great risk). Only the "PlaySmart Full Game" arm (n=3) was asked perception of risk of harm questions at baseline and post gameplay. Qualitative focus group feedback was collected from all other arms.
  units on a scale
    number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    (all) | 2.8 [1.6 to 3.4] |  |  |  |  |  |  |  |  | 2.8 [1.6 to 3.4]

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Questions
Description: Participants were asked 5 true/false knowledge questions pre/post gameplay.
Time Frame: Post Gameplay, up to 1 week
Population: Only 3 participants played the full game.
Measure: Mean (Standard Deviation); unit: Percentage of Questions Correct
Arm/Group | PlaySmart Full Game
Number analyzed (Participants) | 3
Percentage of Questions Correct | 100 (0)

2. Primary Outcome: Perception of Risk of Harm
Description: Participants were asked 5 perception of harm questions then asked to rate the questions on a 4-point scale (no risk to great risk). Change in perception of risk of harm pre/post gameplay was measured to assess this outcome.
Time Frame: Post Gameplay, up to 1 week
Population: Only 3 participants played the full game
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | PlaySmart Full Game
Number analyzed (Participants) | 3
score on a scale | 1 [0 to 3]

3. Primary Outcome: Gameplay Experience
Description: Gameplay experience was assessed using 8 statements to be rated on a scale of 1-5 (1= Not at all, 5= A lot) such as "I was absorbed in this experience" and "I understood the stories in PlaySmart." Each item was assessed individually to assess gameplay experience.
Time Frame: Post Gameplay, up to 1 week
Population: Only 3 participants played the full game.
Measure: Mean (Full Range); unit: Rating on a Scale
Arm/Group | PlaySmart Full Game
Number analyzed (Participants) | 3
Rating on a Scale
  I felt like I was in control of the game. | 3.33 [2 to 5]
  I felt frustrated while playing PlaySmart. | 2.67 [2 to 3]
  I found PlaySmart confusing to use. | 2 [2 to 2]
  I liked the art and design of PlaySmart. | 4.67 [4 to 5]
  I understood the stories in PlaySmart. | 3 [2 to 4]
  I was absorbed in the experience. | 3.33 [3 to 4]
  Playing PlaySmart was interesting. | 4 [4 to 4]
  This game helped me. | 3.67 [3 to 4]

4. Primary Outcome: Beta Test a Storyline of PlaySmart Game
Description: Each storyline was randomly tested by 4 users and they provided qualitative feedback during focus groups post gameplay. Presented are counts of participants that successfully completed this task.
Time Frame: Post Gameplay, up to 1.5 hour
Population: Included are participants who did not play the full game.
Measure: Count of Participants; unit: Participants
Arm/Group | Trading Wisdom Storyline | Lean on Me Storyline | Tough Love Storyline | Grandma's Pills Storyline | A Friend in Need Storyline | A New Direction Storyline
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
Participants | 4 | 4 | 4 | 4 | 4 | 4

5. Primary Outcome: Beta Test PlaySmart Risk Sense Mini Game
Description: Each level of the Risk Sense mini game was randomly tested by 3 users and they provided qualitative feedback during focus groups post gameplay. Presented are counts of participants that successfully completed this task.
Time Frame: Post Gameplay, up to 1.5 hour
Population: 3 participants were randomly selected
Measure: Count of Participants; unit: Participants
Arm/Group | Risk Sense All Levels
Number analyzed (Participants) | 3
Participants | 3

6. Primary Outcome: Beta Test PlaySmart Full Game: Character Development Focus
Description: The PlaySmart Full Game was randomly tested by 3 users and they provided qualitative feedback during focus groups post gameplay focused on character development. Presented are counts of participants that successfully completed the task.
Time Frame: Post Gameplay, up to 1 week
Population: 3 participants were randomly selected
Measure: Count of Participants; unit: Participants
Arm/Group | PlaySmart Full Game: Focus on Character Development
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | PlaySmart Full Game | Trading Wisdom Storyline | Lean on Me Storyline | Tough Love Storyline | Grandma's Pills Storyline | A Friend in Need Storyline | A New Direction Storyline | Risk Sense All Levels | PlaySmart Full Game: Focus on Character Development
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04109599/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04109599/ICF_001.pdf